CLINICAL TRIAL: NCT06969404
Title: Prognostic Value of Capillary Lactatemia in Potentially Severe Polytrauma in Pre-hospital Care
Brief Title: Prognostic Value of Capillary Lactatemia in Potentially Severe Polytrauma Patients
Acronym: CLAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-AOI-05
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- polytrauma patient (Other): capillary blood sampling
  Interventions: Biological: capillary blood sampling

INTERVENTIONS:
Biological: capillary blood sampling — capillary blood sampling during the hospital transfert

SUMMARY:
Nowadays, the tools available to assess the severity of a polytrauma patient in the pre-hospital setting (vital parameters, shock index, MGAP score, Vittel criteria) have their limitations and are sometimes subjective. To date, there are no objective, practical and reproducible tools for triaging these patients. Venous lactataemia also appears to be predictive of poor outcome in severe trauma. However, there are no studies in the literature on capillary lactataemia, which would indicate the potential severity of a polytrauma patient in the pre-hospital setting. However, it is an easily performed, risk-free assay, the results of which can be obtained rapidly at the scene of the accident. The aim of this project is to confirm that, like venous lactataemia, capillary lactataemia can be useful in the pre-hospital phase for predicting a patient's poor outcome. Incorporating this assay into the assessment of potentially severe polytrauma patients in the pre-hospital phase could improve the predictive value of clinical and contextual data and thus enable better referral and management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Presenting a potentially serious pre-hospital trauma defined by:

  o A road accident or a fall of more than 2 metres
* Requiring the dispatch of a SMUR 06 team (mobile emergency and resuscitation service)
* And transferred to an emergency facility in the Alpes Maritimes with medical assistance.
* Consent signed (by the patient or a relative) after the event if it is not possible to sign immediately.
* Pregnant women may also take part in the study without any risk to themselves or their child.

Exclusion Criteria:

* Patients with isolated peripheral limb trauma (wrist, elbow, knee, ankle, shoulder)
* Patients under legal protection (guardianship, curatorship)
* Patients in cardiorespiratory arrest when taken into care by the SMUR (emergency medical services)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
lactemie value H0 | at inclusion
  dosage of capillary lactemia in mmol/L
lactemie value H6 | 6 hours
  dosage of capillary lactemia in mmol/L

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Antibes Hospital, Antibes
  - Cannes hospital, Cannes
  - Nice University Hospital, Nice

IPD SHARING:
Plan to Share IPD: No